CLINICAL TRIAL: NCT06086496
Title: Evaluation of Effectiveness and Safety of Abluminal Biodegradable Polymer Sirolimus-eluting Stent in Routine Clinical Practice: A Prospective, Single-arm, Multicenter, Observational Study (The GENCOMX Registry)
Brief Title: Effectiveness and Safety of Abluminal Biodegradable Polymer Sirolimus-eluting Stent (GENOSS® DES)
Acronym: GENCOMX
Status: Enrolling by invitation | Type: Observational
Sponsor: Genoss Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2022AN0320
Record Dates: First submitted 2023-10-04; First posted 2023-10-17 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Coronary Artery Disease; Percutaneous Coronary Intervention
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- GENOSS® DES Sirolimus Eluting Coronary Stent System / B03300.20, class [4]: Patients with coronary artery disease who require interventional treatment through stent insertion in real-world practice (all-comer)
  Interventions: Device: GENOSS® DES Sirolimus Eluting Coronary Stent System

INTERVENTIONS:
Device: GENOSS® DES Sirolimus Eluting Coronary Stent System — The GENOSS® DES is L-605 cobalt chromium (CoCr) platform with a strut thickness of 70µm Sirolimus drug with concentration of 1.15µg/mm2 Abluminal biodegradable PLA and PLGA polymers.

SUMMARY:
In this study, the investigators evaluated the effectiveness and safety of using the GENOSS® DES, which has a biodegradable polymer only on the inner wall of the blood vessel, for patients(all-comers) with coronary artery disease who require percutaneous coronary intervention through stent insertion.

DETAILED DESCRIPTION:
This study is a sponsor-initiated clinical trial (SIT) that enrolls patients who underwent percutaneous coronary intervention using the GENOSS® DES drug-eluting stent.

As it is a prospective, multicenter, observational study, the number of subjects is not separately calculated, but the plan is to recruit a total of 1,000 participants at 7 institutions during the study registration period.

ELIGIBILITY:
<Inclusion Criteria>

1. Adults over 19 years of age
2. Patients with typical symptoms or objective evidence of myocardial ischemia and eligible for coronary angioplasty.
3. Severe coronary artery stenosis suitable for GENOSS® DES insertion
4. Patients who agree to the research protocol and clinical follow-up plan and give written informed consent in the consent form approved by the Institutional Review Board/Ethics Committee of each research institution.

<Exclusion Criteria>

1. Test subjects with known hypersensitivity or contraindications to the following drugs or substances: heparin, aspirin, clopidogrel, sirolimus, contrast medium (however, even subjects with hypersensitivity to contrast medium can be controlled by steroids and pheniramine) In this case, registration is possible, but if there is known anaphylaxis, it is excluded)
2. Patients who also received other drug-eluting stents
3. If you have a disease with a remaining life expectancy of less than 1 year
4. Pregnant or lactating women or women who may be pregnant
5. Cases in which the patient was admitted to the hospital due to psychogenic shock and the likelihood of survival is medically expected to be low.
6. Patients judged by researchers to be unsuitable for research

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Coronary artery disease patients who underwent coronary intervention using the GENOSS® DES
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Target Lesion Failure (TLF) | at 12 months after the procedure
  The composite end point of cardiac death, TV-MI (target vessel-MI), and TLR (target lesion revascularization)

SECONDARY OUTCOMES:
All deaths | at 12 months after the procedure
Cardiac death | at 12 months after the procedure
TV-MI (target vessel-myocardial infarction) | at 12 months after the procedure
any MI (myocardial infarction) | at 12 months after the procedure
ID-TVR (ischemia-driven target vessel revascularization) | at 12 months after the procedure
ID-TLR (ischemia-driven target lesion revascularization) | at 12 months after the procedure
Stent thrombosis by ARC definition | at 12 months after the procedure
Procedure success | during the hospitalization period (up to 3 days)
  When the final internal stenosis rate is less than 30% as assessed visually on angiography after the procedure and there is no death, Q-wave myocardial infarction, or urgent revascularization during hospitalization.

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Anam Hospital, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
The data set is available from the the corresponding author upon reasonable request.